CLINICAL TRIAL: NCT00397774
Title: Phase 3 Physical Activity and Functioning in Palliative Cancer Patients - a Clinical Randomised Trial
Brief Title: Physical Activity and Functioning in Palliative Cancer Patients - a Clinical Randomised Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4.2006.2179
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Cancer
Keywords: Palliative care; Physical exercise; Physical function
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Active Comparator): Physical exercise twice a week for 8 weeks, and best supportive care
  Interventions: Behavioral: Physical exercise; Other: best supportive care
- No exercise (Other): Best supportive care, no exercise
  Interventions: Other: best supportive care

INTERVENTIONS:
Behavioral: Physical exercise — Physical exercise twice a week for 8 weeks, and best supportive care
  Arms: Exercise
Other: best supportive care

SUMMARY:
The project consists of two studies where we want to throw light on the importance of physical activity/exercise to maintain physical function among cancer patients whose disease is not responsive to curative treatment. Study I is a randomised intervention study where we want to study the effect of adjusted physical exercise compared to usual care. In study II our main aim is to validate different subjective and objective methods to measure physical functioning

ELIGIBILITY:
Inclusion Criteria:

* Palliative cancer patients,
* life expectancy between 3 and 12 months,
* Karnofsky status equally or above 60,
* pain score equal or below 3 on numerical rating scale (0-10),
* cognitive function intact

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2006-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Fatigue | immediately before and after the intervention

SECONDARY OUTCOMES:
Health related quality of life and physical functioning | immediately before and after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Line M Oldervoll, PhD, Principal Investigator — Department of Cancer Reserach and Molecular Medicine
Locations (5):
- Norway (5):
  - Sunniva Clinic for Palliative Care, Bergen
  - Hospice Lovisenberg, Oslo
  - Oslo University Hospital, Oslo
  - Telemark Hospital, Skien
  - St. Olavs University Hospital, Trondheim

REFERENCES:
- [Result] Oldervoll LM, Loge JH, Lydersen S, Paltiel H, Asp MB, Nygaard UV, Oredalen E, Frantzen TL, Lesteberg I, Amundsen L, Hjermstad MJ, Haugen DF, Paulsen O, Kaasa S. Physical exercise for cancer patients with advanced disease: a randomized controlled trial. Oncologist. 2011;16(11):1649-57. doi: 10.1634/theoncologist.2011-0133. Epub 2011 Sep 26. PMID 21948693